CLINICAL TRIAL: NCT02229552
Title: Habituation to Food as a Risk Factor for Pediatric Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Leonard Epstein, Principal Investigator, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 1102924-1-61250
Record Dates: First submitted 2014-07-18; First posted 2014-09-01 (Estimated); Results first posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Obesity in Children
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Children completed measurements of body weight, habituation to food, questionnaires and cognitive assessments in a repeated assessment prospective study.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Baseline Cohort (Other): Children completed body weight and other measures at baseline, 1-year follow up and 2-year follow up measurement periods.
  Interventions: Other: Standardized Assessments

INTERVENTIONS:
Other: Standardized Assessments — Children were asked to attend appointments without consuming study foods 24 hours previously, as habituation measurements are sensitive to recent consumption. Children were provided access to snack prior to completing questionnaires or cognitive assessments. Habituation to food, questionnaires and cognitive assessments were re-measured at 1-year and 2-year follow up.

SUMMARY:
The study is designed to assess habituation of behavioral responding for food as risk factors for increases in Standardized Body Mass Index (zBMI) over two years in non-overweight children.

DETAILED DESCRIPTION:
Cross sectional data have shown slower habituation is related to greater energy intake, and habituation is slower for overweight/obese compared to leaner youth, but it is not known whether this is a result of being overweight, or whether slower habituation is a risk factor for weight gain. The goal of this application is to study individual differences in behavioral (responding for food) habituation as risk factors for alterations in zBMI and body fat over a two year period in 200, 8 to 12 year-old non-overweight children. This project will provide the first test of the hypothesis that slow habituation to food is a risk factor for increases in zBMI in non-overweight youth.

ELIGIBILITY:
Inclusion Criteria:

* 8-12 years of age
* Participants will include children who are at the 50th BMI percentile and less than the 85th BMI percentile (BMI = kg/m2) at baseline. We will also include children who are below the 50th percentile, but have at least one biological parent with a current BMI ≥ 25 kg/m2.

Exclusion Criteria:

* Food allergies or special diets: Youth should have no dietary restrictions that could interfere with these experiments, including food allergies or religious or ethnic practices that limit food choice or medical conditions which alter nutritional status or intestinal absorption (e.g. inflammatory bowel disease).
* Activity restrictions: Children who have activity restrictions due to medical or physical problems, such as uncontrolled exercise induced asthma or a disability requiring wheelchair use will not participate.
* Psychopathology, medications or sickness: Children should have no psychopathology (e.g. childhood schizophrenia) or developmental disabilities that would limit participation. Children will also be excluded if they are taking medications that could affect their level of activity or appetite (e.g. methylphenidate).
* Moderate or greater liking of study foods. Children must report at least a moderate liking ( 3 or greater on a 5-point Likert-type scale) of the foods used in these studies and be willing to consume them.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 237 (Actual)
Dates: Start 2012-11; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Epstein, Ph.D., Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Epstein LH, Carr KA, O'Brien A, Paluch RA, Temple JL. High reinforcing value of food is related to slow habituation to food. Eat Behav. 2020 Aug;38:101414. doi: 10.1016/j.eatbeh.2020.101414. Epub 2020 Jul 29. PMID 32799072
- [Derived] Epstein LH, Carr KA, Scheid JL, Gebre E, O'Brien A, Paluch RA, Temple JL. Taste and food reinforcement in non-overweight youth. Appetite. 2015 Aug;91:226-32. doi: 10.1016/j.appet.2015.04.050. Epub 2015 Apr 16. PMID 25891040
- [Derived] Kong KL, Feda DM, Eiden RD, Epstein LH. Origins of food reinforcement in infants. Am J Clin Nutr. 2015 Mar;101(3):515-22. doi: 10.3945/ajcn.114.093237. Epub 2015 Jan 14. PMID 25733636
- See also: UB Division of Behavioral Medicine Website — http://medicine.buffalo.edu/departments/pediatrics/divisions/behavioral-medicine.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Baseline Cohort: All children completed the same baseline measures
Period: Baseline
Arm/Group | Baseline Cohort
Started | 237
Completed | 231
Not Completed | 6
Not completed — Withdrawal by Subject | 6
Period: 1-year Follow up
Arm/Group | Baseline Cohort
Started | 231
Completed | 206
Not Completed | 25
Not completed — Withdrawal by Subject | 7
Not completed — Lost to Follow-up | 18
Period: 2-Year Follow up
Arm/Group | Baseline Cohort
Started | 231 (All baseline participants were eligible for year 2 follow up, regardless of completion of year 1.)
Completed | 205
Not Completed | 26
Not completed — Withdrawal by Subject | 9
Not completed — Lost to Follow-up | 17

BASELINE CHARACTERISTICS:
Groups:
- Baseline Cohort: All children completed measures of habituation to food, questionnaires and cognitive assessments at baseline and 1-year and 2-year follow up periods.
Arm/Group | Baseline Cohort
Number analyzed (Participants) | 231
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.45 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120
  Male | 111
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14
  Not Hispanic or Latino | 215
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 33
  White | 170
  More than one race | 22
  Unknown or Not Reported | 2
Height [Mean (Standard Deviation); unit: Centimeters] | 142.89 (11.4)
Weight [Mean (Standard Deviation); unit: pounds] | 78.33 (18.28)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 17.15 (1.77)
Body Composition [Mean (Standard Deviation); unit: Percent body fat] | 16.52 (5.95)
zBMI [Mean (Standard Deviation); unit: z-score BMI] — The BMI Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the population mean, based on age and sex. Negative numbers indicate values lower than the mean and positive numbers indicate values higher than the mean. A lower z-score indicates less obesity, with numbers between -1.0 and +1.0 indicating normal weight and numbers greater than 1.0 indicating an overweight status.
  z-score BMI | -0.039 (0.72)

OUTCOME MEASURES:

1. Primary Outcome: Change in zBMI
Description: To assess the rate of habituation of behavioral responding to savory, sweet and salty foods as independent or interactive risk factors for zBMI trajectories, with the hypothesis that the rate of habituation of behavioral responding for food predicts zBMI trajectories over time, controlling for child gender, parental education, parental BMI, physical activity, ethnicity, the reinforcing value of food and eating in the absence of hunger.
Time Frame: 2 years
Population: 205 children completed baseline, year one height and weight measures and year two follow up height and weight measures
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | Baseline Cohort
Number analyzed (Participants) | 205
z-score
  Baseline Measures | -0.048 (0.744)
  1-year follow up measures | 0.013 (0.759)
  2-year follow up measures | 0.011 (0.807)
Statistical Analysis 1: Comparison: Baseline Cohort; Test type: Other — Repeated measures analysis of variance with zbmi for each year as the repeated dependent measure; p = 0.051, ANOVA; Mean Difference (Final Values) = 3.00

ADVERSE EVENTS:
Time Frame: 2 years
Description: Only participation-related adverse events were collected.
Arm/Group | Baseline Cohort
All-Cause Mortality (participants affected / at risk) | 0/237
Serious Adverse Events (participants affected / at risk) | 0/237
Other Adverse Events (participants affected / at risk) | 0/237

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No